CLINICAL TRIAL: NCT04109313
Title: An Open-label, Multicenter, Extension Study to Evaluate the Long-term Safety and Tolerability of LOU064 in Eligible Subjects With CSU Who Have Participated in CLOU064A2201
Brief Title: An Open-label Extension Study to Evaluate the Long-term Safety and Tolerability of LOU064 in Subjects With CSU
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLOU064A2201E1; 2019-001074-29 (EudraCT Number)
Record Dates: First submitted 2019-09-27; First posted 2019-09-30 (Actual); Results first posted 2023-09-29 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Chronic Spontaneous Urticaria
Keywords: Chronic spontaneous urticaria; BTK Inhibitor; Long term safety; Urticaria activity score
MeSH Terms: conditions — Chronic Urticaria | interventions — remibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- All participants (Experimental): Participants with UAS7<16 at Week 16 of CLOU064A2201 were followed up to 12 weeks without receiving treatment (observational period). If participants relapsed (UAS7≥16 at least once), they were transitioned to the treatment period. Otherwise, they were discontinued from the study.
  Participants with a UAS7≥16 at Week 12 or Week 16 in the CLOU064A2201, as well as participants who experienced a relapse during the 12-week observational period, were administered 100 mg of LOU064 b.i.d. open-label for up to 52 weeks.
  Interventions: Drug: LOU064

INTERVENTIONS:
Drug: LOU064 — Participants with a UAS7≥16 at Week 12 or Week 16 in the CLOU064A2201, as well as participants who experienced a relapse during the 12-week observational period, were administered LOU064 50mg capsules b.i.d. (i.e. two capsules of LOU064 50mg in the morning and two capsules of LOU064 50mg in the evening) from Day 1 up to Week 52 of the Treatment period.

SUMMARY:
The main objective to assess the long-term safety and tolerability of LOU064 in patients with chronic spontaneous urticaria (CSU) who have participated in study CLOU064A2201 (NCT03926611)

DETAILED DESCRIPTION:
This was an open-label, single-arm, multicenter, long-term safety and tolerability extension study for CSU patients rolling over from study CLOU064A2201 (NCT03926611).

Subjects rolling over from CLOU064A2201 with a weekly Urticaria Activity Score (UAS7)<16 after the follow-up period at Week 16 were further followed up without receiving LOU064 for up to 12 weeks (observational period). If there was a relapse (UAS7≥16 at least once), the 12-week observational period was terminated, and subjects entered the treatment period. Subjects who never relapsed within 12 weeks completed the study after the observational period without treatment.

Subjects who rolled over from CLOU064A2201 with a UAS7≥16 at Week 12 or Week 16, as well as those subjects who relapsed during the 12-week observational period, were treated with 100 mg LOU064 twice a day (b.i.d.) open-label for 52 weeks. No background medication with a second-generation H1-antihistamine was permitted up to Week 4 of the treatment period. Subjects who completed the treatment period or who discontinued treatment early were followed-up for a minimum duration of 4 weeks. Subjects who had a UAS7≤6 at Week 52 of the treatment period had their follow-up period extended until relapse (UAS7≥16) for up to a total of 16 weeks.

ELIGIBILITY:
Key Inclusion Criteria:

* Participants must provide written informed consent prior to any assessments.
* Participants must be willing and able to complete a daily symptom eDiary throughout the study and adhere to the study visit schedules.
* Participants transitioning from the CLOU064A2201 trial must have completed either the Week 12 visit (end of treatment period) or the Week 16 visit (end of follow-up period). They will be assigned to either the treatment period or the observational period based on their UAS7 score (average score from the 7 days prior to the respective visit) as follows:

  1. Participants transitioning at Week 12 of CLOU064A2201 with a UAS7 score of ≥16 will be allocated to the treatment period.
  2. Participants transitioning at Week 16 of CLOU064A2201 with a UAS7 score of ≥16 will be allocated to the treatment period.
  3. Participants transitioning at Week 16 of CLOU064A2201 with a UAS7 score of <16 will be allocated to the observational period.

Key Exclusion Criteria:

* Participants with a clearly defined predominant or sole trigger for their chronic urticaria, such as chronic inducible urticaria (including symptomatic dermographism, cold-induced, heat-induced, solar-induced, pressure-induced, delayed pressure-induced, aquagenic-induced, cholinergic-induced, or contact-induced urticaria).
* Participants with other diseases presenting with urticaria or angioedema symptoms, including but not limited to urticaria vasculitis, urticarial pigmentosa, erythema multiforme, mastocytosis, hereditary urticaria, or acquired/drug-induced urticaria.
* Participants with any other skin disease associated with chronic itching that, in the opinion of the investigator, could affect the study evaluations and results, such as atopic dermatitis, bullous pemphigoid, dermatitis herpetiformis, senile pruritus, or psoriasis.
* Participants with a history or current diagnosis of ECG abnormalities that indicate a significant safety risk for their participation in the study, including:
* Concomitant clinically significant cardiac arrhythmias (e.g., sustained ventricular tachycardia) and clinically significant second or third-degree AV block without a pacemaker.
* History of familiar long QT syndrome or a known family history of Torsades de Pointes.
* Resting heart rate (as determined by physical exam or 12-lead ECG) below 50 bpm.
* Resting QTcF interval ≥450 msec (in males) or ≥460 msec (in females) at day 1 of the treatment period or inability to determine the QTcF interval.
* Use of agents known to prolong the QT interval, unless they can be permanently discontinued for the duration of the study.
* Participants with a significant risk of bleeding or coagulation disorders.
* Participants with a known or suspected history of an ongoing, chronic, or recurrent infectious disease, including but not limited to opportunistic infections (e.g., tuberculosis, atypical mycobacterioses, listeriosis, or aspergillosis), HIV, or Hepatitis B/C.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2019-10-24 (Actual); Primary Completion 2022-09-09 (Actual); Study Completion 2022-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceutical, Study Director — Novartis Pharmaceutical
Locations (62):
- United States (10):
  - Novartis Investigative Site, Litchfield Park, Arizona
  - Novartis Investigative Site, Little Rock, Arkansas
  - Novartis Investigative Site, Mission Viejo, California
  - Novartis Investigative Site, San Diego, California
  - Novartis Investigative Site, Walnut Creek, California
  - Novartis Investigative Site, Pembroke Pines, Florida
  - Novartis Investigative Site, Owensboro, Kentucky
  - Novartis Investigative Site, Ypsilanti, Michigan
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Grove City, Ohio
- Argentina (4):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, La Plata, Buenos Aires
  - Novartis Investigative Site, Mendoza, Mendoza Province
  - Novartis Investigative Site, CABA
- Belgium (2):
  - Novartis Investigative Site, Edegem, Antwerpen
  - Novartis Investigative Site, Liège
- Canada (6):
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, London, Ontario
  - Novartis Investigative Site, Niagara Falls, Ontario
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Québec, Quebec
  - Novartis Investigative Site, Verdun, Quebec
- Czechia (3):
  - Novartis Investigative Site, Prague, Czech Republic
  - Novartis Investigative Site, Prague, Prague 1
  - Novartis Investigative Site, Tábor
- Denmark (2):
  - Novartis Investigative Site, Arhus C
  - Novartis Investigative Site, Copenhagen NV
- France (3):
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Nice
- Hungary (5):
  - Novartis Investigative Site, Orosháza, Bekes County
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Pécs
  - Novartis Investigative Site, Szolnok
- Japan (7):
  - Novartis Investigative Site, Ichinomiya, Aichi-ken
  - Novartis Investigative Site, Funabashi, Chiba
  - Novartis Investigative Site, Hiroshima, Hiroshima
  - Novartis Investigative Site, Obihiro, Hokkaido
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Itabashi-ku, Tokyo
  - Novartis Investigative Site, Takaoka, Toyama
- Poland (4):
  - Novartis Investigative Site, Gdansk
  - Novartis Investigative Site, Lodz
  - Novartis Investigative Site, Rzeszów
  - Novartis Investigative Site, Warsaw
- Russia (3):
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Stavropol
- Slovakia (3):
  - Novartis Investigative Site, Košice, Slovak Republic
  - Novartis Investigative Site, Nové Zámky
  - Novartis Investigative Site, Svidník
- Spain (3):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Alicante, Valencia
  - Novartis Investigative Site, Madrid
- Turkey (Türkiye) (3):
  - Novartis Investigative Site, Istanbul, TUR
  - Novartis Investigative Site, Denizli
  - Novartis Investigative Site, Talas / Kayseri
- United Kingdom (4):
  - Novartis Investigative Site, Leeds
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Oxford
  - Novartis Investigative Site, Plymouth

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing access to patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to protect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Jain V, Gimenez-Arnau A, Hayama K, Reich A, Carr W, Tillinghast J, Dahale S, Lheritier K, Walsh P, Zharkov A, Hugot S, Haemmerle S. Remibrutinib demonstrates favorable safety profile and sustained efficacy in chronic spontaneous urticaria over 52 weeks. J Allergy Clin Immunol. 2024 Feb;153(2):479-486.e4. doi: 10.1016/j.jaci.2023.10.007. Epub 2023 Oct 20. PMID 37866460
- See also: Patient Lay Trial Summary — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1569

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 229 subjects were enrolled in the observational period or the treatment period across 72 sites in 15 countries.
  One subject was a screening failure and, as a result, was not enrolled in either the observational or treatment period.
Pre-assignment Details: Participants with UAS7<16 at Week 16 of CLOU064A2201 (NCT03926611) entered a 12-week observational period.
  Participants with UAS7≥16 at Week 12 or Week 16 of CLOU064A2201, as well as those who relapsed during the observational period, entered the treatment period.
Groups:
- All Participants: Participants with UAS7<16 at Week 16 of CLOU064A2201 were followed up to 12 weeks without receiving treatment (observational period). If participants relapsed (UAS7≥16 at least once), they were transitioned to the treatment period.
  Participants with a UAS7≥16 at Week 12 or Week 16 in the CLOU064A2201, as well as participants who experienced a relapse during the 12-week observational period, were administered 100 mg of LOU064 b.i.d. open-label for up to 52 weeks.
Period: Overall Study
Arm/Group | All Participants
Started | 229
Treatment-free Cohort (Participants with UAS7<16 at Week 16 of CLOU064A2201 were followed up to 12 weeks without receiving treatment (observational period). If participants relapsed (UAS7≥16 at least once), they were transitioned to the treatment period. Otherwise, the) | 68
Treatment Cohort (Participants with a UAS7≥16 at Week 12 or Week 16 in the CLOU064A2201, as well as participants who experienced a relapse during the 12-week observational period, were administered 100 mg of LOU064 b.i.d. open-label for up to 52 weeks.) | 194
Completed | 188
Not Completed | 41
Not completed — Pregnancy | 1
Not completed — Adverse Event | 11
Not completed — Lack of Efficacy | 11
Not completed — Lost to Follow-up | 1
Not completed — Physician Decision | 2
Not completed — Subject Decision | 13
Not completed — Covid-19 situation | 2

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 229
Age, Continuous [Median (Full Range); unit: Years] | 45 [18 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 165
  Male | 64
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 181
  Black | 2
  Asian | 44
  Multiple | 1
  American Indian or Alaska Native | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (AEs)
Description: An AE refers to any undesirable medical occurrence, such as an unintended sign (including abnormal laboratory findings), symptom, or disease, experienced by a participant. Serious AEs (SAEs) is defined as any AE that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, results in a congenital anomaly/birth defect, or any other medically significant condition.
  Treatment-emergent AEs were defined as AEs that either begin on the same day or after the first dose of study medication during the treatment period in the extension study or worsen on the same day or after the first dose of study medication in the extension study and within the minimum of either 28 days post last dose or the end of the study visit. The number of participants with treatment-emergent AEs was summarized.
Time Frame: From first dose of treatment up to 28 days after last dose, assessed up to 56 weeks
Population: All subjects who received at least one dose of study treatment during the treatment period of this extension study.
Measure: Count of Participants; unit: Participants
Groups:
- Treated Cohort: Participants with a UAS7≥16 at Week 12 or Week 16 in the CLOU064A2201, as well as participants who experienced a relapse during the 12-week observational period, were administered 100 mg of LOU064 b.i.d. open-label for up to 52 weeks.
Arm/Group | Treated Cohort
Number analyzed (Participants) | 194
Participants
  AEs | 139
  Deaths | 0
  Non-fatal Serious AEs (SAEs) | 6
  SAE(s) | 6
  Discontinued treatment due to any AE(s) | 11
  Discontinued treatment due to any SAE(s) | 2
  Treatment interruption due to AE(s) | 13
  Treatment interruption due to SAE(s) | 1

2. Secondary Outcome: Change From Baseline in Weekly Urticaria Activity Score (UAS7) at Week 4 of the Treatment Period
Description: The Urticaria Activity Score (UAS) is a composite, diary-recorded score with numeric severity intensity ratings (0=none to 3=intense/severe) for the number of wheals (hives) and the intensity of the pruritus (itch) over the past 12 hours (twice daily). The daily UAS is calculated as the average of the morning and evening scores. The UAS7 is the weekly sum of the daily UAS, which is the composite score of the intensity of pruritus and the number of wheals. UAS7 scores ranged from 0 to 42. A higher UAS7 indicated greater urticaria disease activity. A minimum of 4 out of 7 daily scores were needed to calculate the UAS7 values. Otherwise, the weekly score was missing for that week.
  The change from baseline in UAS7 at Week 4 of the treatment period was calculated. A negative change score from baseline indicates improvement. The UAS7 at baseline was considered as the UAS7 derived over the last 7 days before day 1 of the treatment period.
Time Frame: Baseline, Week 4 of treatment period
Population: All subjects who received at least one dose of study treatment during the treatment period of this extension study with a value at both baseline and Week 4 of the treatment period.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Treated Cohort
Number analyzed (Participants) | 187
Score on a Scale | -17.58 (13.400)

3. Secondary Outcome: Percentage of Participants With Well-controlled Disease (UAS7≤6) at Week 4 of the Treatment Period
Description: The Urticaria Activity Score (UAS) is a composite, diary-recorded score with numeric severity intensity ratings (0=none to 3=intense/severe) for the number of wheals (hives) and the intensity of the pruritus (itch) over the past 12 hours (twice daily). The daily UAS is calculated as the average of the morning and evening scores. The UAS7 is the weekly sum of the daily UAS, which is the composite score of the intensity of pruritus and the number of wheals. UAS7 scores ranged from 0 to 42. A higher UAS7 indicated greater urticaria disease activity.
  A minimum of 4 out of 7 daily scores were needed to calculate the UAS7 values. Otherwise, the weekly score was missing for that week. Missing values were imputed by non-responder imputation method regardless of the reason for missingness.
  The percentage of subjects with UAS7≤ 6 at Week 4 of the treatment period was calculated. The 90% confidence interval was derived based on the score method with continuity correction.
Time Frame: Week 4 of the treatment period
Population: All subjects who received at least one dose of study treatment during the treatment period of this extension study.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Treated Cohort
Number analyzed (Participants) | 194
Percentage of participants | 51.0 [44.9 to 57.1]

4. Secondary Outcome: Percentage of Participants With Complete Response (UAS7=0) at Week 4 of the Treatment Period
Description: The Urticaria Activity Score (UAS) is a composite, diary-recorded score with numeric severity intensity ratings (0=none to 3=intense/severe) for the number of wheals (hives) and the intensity of the pruritus (itch) over the past 12 hours (twice daily). The daily UAS is calculated as the average of the morning and evening scores. The UAS7 is the weekly sum of the daily UAS, which is the composite score of the intensity of pruritus and the number of wheals. UAS7 scores ranged from 0 to 42. A higher UAS7 indicated greater urticaria disease activity.
  A minimum of 4 out of 7 daily scores were needed to calculate the UAS7 values. Otherwise, the weekly score was missing for that week. Missing values were imputed by non-responder imputation method regardless of the reason for missingness.
  The percentage of subjects with UAS7= 0 at Week 4 of the treatment period was calculated. The 90% confidence interval was derived based on the score method with continuity correction.
Time Frame: Week 4 of the treatment period
Population: All subjects who received at least one dose of study treatment during the treatment period of this extension study.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Treated Cohort
Number analyzed (Participants) | 194
Percentage of participants | 27.3 [22.2 to 33.1]

5. Secondary Outcome: Percentage of Participants With Well-controlled Disease (UAS7≤ 6) Overtime
Description: The Urticaria Activity Score (UAS) is a composite, diary-recorded score with numeric severity intensity ratings (0=none to 3=intense/severe) for the number of wheals (hives) and the intensity of the pruritus (itch) over the past 12 hours (twice daily). The daily UAS is calculated as the average of the morning and evening scores. The UAS7 is the weekly sum of the daily UAS, which is the composite score of the intensity of pruritus and the number of wheals. UAS7 scores ranged from 0 to 42. A higher UAS7 indicated greater urticaria disease activity.
  A minimum of 4 out of 7 daily scores were needed to calculate the UAS7 values. Otherwise, the weekly score was missing for that week.
  The percentage of subjects with UAS7≤ 6 during the treatment period was calculated. The 90% confidence interval was derived based on the score method with continuity correction. The UAS7 at baseline was considered as the UAS7 derived over the last 7 days before day 1 of the treatment period.
Time Frame: From baseline until Week 52 of the treatment period
Population: All subjects who received at least one dose of study treatment during the treatment period of this extension study. Number analyzed refers to the number of participants with an evaluable value at the specified time points.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Treated Cohort
Number analyzed (Participants) | 194
Percentage of participants
  Baseline: number analyzed (Participants) | 193
  Baseline | 1.0 [0.2 to 3.5]
  Week 1: number analyzed (Participants) | 179
  Week 1 | 37.4 [31.4 to 43.8]
  Week 4: number analyzed (Participants) | 188
  Week 4 | 52.7 [46.4 to 58.8]
  Week 12: number analyzed (Participants) | 173
  Week 12 | 56.6 [50.1 to 63.0]
  Week 20: number analyzed (Participants) | 169
  Week 20 | 62.7 [56.1 to 68.9]
  Week 28: number analyzed (Participants) | 162
  Week 28 | 68.5 [61.9 to 74.5]
  Week 40: number analyzed (Participants) | 155
  Week 40 | 66.5 [59.6 to 72.7]
  Week 52: number analyzed (Participants) | 147
  Week 52 | 68.0 [61.1 to 74.3]

6. Secondary Outcome: Change From Baseline in UAS7 Overtime
Description: The Urticaria Activity Score (UAS) is a composite, diary-recorded score with numeric severity intensity ratings (0=none to 3=intense/severe) for the number of wheals (hives) and the intensity of the pruritus (itch) over the past 12 hours (twice daily). The daily UAS is calculated as the average of the morning and evening scores. The UAS7 is the weekly sum of the daily UAS, which is the composite score of the intensity of pruritus and the number of wheals. UAS7 scores ranged from 0 to 42. A higher UAS7 indicated greater urticaria disease activity.
  A minimum of 4 out of 7 daily scores were needed to calculate the UAS7 values. Otherwise, the weekly score was missing for that week.
  The change from baseline in UAS7 during the treatment period was calculated. A negative change score from baseline indicates improvement. The UAS7 at baseline was considered as the UAS7 derived over the last 7 days before day 1 of the treatment period.
Time Frame: From baseline until Week 52 of the treatment period
Population: Subjects who received at least one dose of study treatment during the treatment period of this extension study and did not have missing values at the specified time points. Number analyzed refers to the number of participants with an evaluable value at the specified time points.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Treated Cohort
Number analyzed (Participants) | 193
Score on a Scale
  Week 1: number analyzed (Participants) | 178
  Week 1 | -14.76 (11.502)
  Week 4: number analyzed (Participants) | 187
  Week 4 | -17.58 (13.400)
  Week 12: number analyzed (Participants) | 172
  Week 12 | -19.37 (12.502)
  Week 20: number analyzed (Participants) | 168
  Week 20 | -20.61 (11.634)
  Week 28: number analyzed (Participants) | 161
  Week 28 | -21.54 (11.525)
  Week 40: number analyzed (Participants) | 154
  Week 40 | -21.25 (11.400)
  Week 52: number analyzed (Participants) | 146
  Week 52 | -21.82 (10.699)

ADVERSE EVENTS:
Time Frame: In the Treated cohort, treatment-emergent AEs were collected from first dose of treatment up to 28 days post last dose, up to 56 weeks; and deaths were collected from first dose of treatment until end of study, assessed up to 68 weeks. In the Treatment-free cohort, AEs and deaths were collected from start of observation period until relapse (UAS7≥16) or end of observation period, up to 12 weeks.
Description: An AE refers to any undesirable medical occurrence, such as an unintended sign (including abnormal laboratory findings), symptom, or disease, experienced by a participant.
Groups:
- Treatment-free Cohort (Observational Period): Participants with UAS7<16 at Week 16 of CLOU064A2201 were followed up to 12 weeks without receiving treatment (observational period). If participants relapsed (UAS7≥16 at least once), they were transitioned to the treatment period (treated cohort).
- Treated Cohort (Treatment+Follow-up Period): Participants with a UAS7≥16 at Week 12 or Week 16 in the CLOU064A2201, as well as participants who experienced a relapse during the 12-week observational period, were administered 100 mg of LOU064 b.i.d. open-label for up to 52 weeks.
Arm/Group | Treatment-free Cohort (Observational Period) | Treated Cohort (Treatment+Follow-up Period)
All-Cause Mortality (participants affected / at risk) | 0/68 | 0/194
Serious Adverse Events (participants affected / at risk) | 1/68 | 6/194
Other Adverse Events (participants affected / at risk) | 0/68 | 56/194
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment-free Cohort (Observational Period) (N=68) | Treated Cohort (Treatment+Follow-up Period) (N=194)
Melaena (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
COVID-19 pneumonia (Infections and infestations) | 0 | 2
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1
Superficial spreading melanoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment-free Cohort (Observational Period) (N=68) | Treated Cohort (Treatment+Follow-up Period) (N=194)
COVID-19 (Infections and infestations) | NA | 16
Headache (Nervous system disorders) | NA | 13
Chronic spontaneous urticaria (Skin and subcutaneous tissue disorders) | NA | 22
Eczema (Skin and subcutaneous tissue disorders) | NA | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-09-08): https://cdn.clinicaltrials.gov/large-docs/13/NCT04109313/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-13): https://cdn.clinicaltrials.gov/large-docs/13/NCT04109313/SAP_001.pdf